CLINICAL TRIAL: NCT06584487
Title: Proximal Metatarsal Medial Opening Wedge Osteotomy Fixed by Plate and Screws in Correction of Hallux Valgus
Brief Title: Proximal Metatarsal Osteotomy in Correction of Hallux Valgus
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdulrahman Mahdi Hussein Mohamed, Resident, Assiut University
Other Study IDs: Hallux valgus osteotomy
Record Dates: First submitted 2024-08-14; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Hallux Valgus and Bunion
Keywords: Proximal Osteotomy; Medial Opening Wedge; Hallux Valgus
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The outcomes of the correction of hallux valgus by proximal opening wedge osteotomy

DETAILED DESCRIPTION:
Hallux valgus is a common cause of foot pain and deformity in the adult and adolescent population, which often requires surgical treatment when nonsurgical treatments fail.

During the past decades, multiple modified procedures and fixation techniques have been described.

The most common types of osteotomies of the first metatarsal are crescentic, chevron, scarf and lateral or medial opening wedge techniques.

A concern with the Chevron and other distal osteotomies is the development of avascular necrosis of the first metatarsal head with a reported incidence of between 0% and 20%.

On the other side, the proximal dome osteotomy along with a distal soft tissue release is an excellent procedure. The proximal location of the osteotomy avoids devascularization of the metatarsal head, and the crescent shape maintains the length of the metatarsal. It allows a high degree of correction at the intermetatarsal angle in severe deformities.

When the condition is associated with an increased intermetatarsal angle, a surgical technique using a proximal first metatarsal osteotomy is often indicated. A proximal opening wedge osteotomy stabilized with a wedge and plate configuration offers a stable, reliable means to correct the increased intermetatarsal angle.

Over the past 10 years, some surgeons have increasingly used locking plates instead of a single screw for stabilisation of the osteotomy with the assumption of better postoperative stability and preserved length of the first metatarsal. In addition, fixation with a plate has been described as technically less challenging.

ELIGIBILITY:
Inclusion Criteria:

* all admitted patients to Assiut University Hospitals.
* age group of 15 years old and above.
* Moderate and severe degrees of hallux valgus.

Exclusion Criteria:

* Burn
* age group below 15 years old.
* patient who refuse to participate in the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patient above 15 years old
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The American Orthopedic Foot and Ankle Society hallux-metatarsophalangeal-interphalangeal scale (AOFAS scale). | baseline
  Pain-Function-Alignment

SECONDARY OUTCOMES:
Post operative radiographic changes in standing AP view foot and standing lateral view foot. | Baseline
  In standing AP view foot
  * The hallux valgus angle HVA in degrees.It is the angle between long axis of 1st metatarsal and proximal phalanx of big toe
  * The intermetatarsal angle IMA in degree
  * The distal metatarsal articular angle DMAA in degree
  * The 1st metatarsal length in centimeter In standing lateral view foot
  * The inclination angle of the 1st metatarsal in degree In standing AP view foot
  * The hallux valgus angle HVA in degree
  * The intermetatarsal angle IMA in degree
  * The distal metatarsal articular angle DMAA in degree
  * The 1st metatarsal length in centimeter In standing lateral view foot
  * The inclination angle of the 1st metatarsal

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman M Hussein Mohamed, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Markbreiter LA, Thompson FM. Proximal metatarsal osteotomy in hallux valgus correction: a comparison of crescentic and chevron procedures. Foot Ankle Int. 1997 Feb;18(2):71-6. doi: 10.1177/107110079701800205. PMID 9043877
- [Background] Saragas NP. Proximal opening-wedge osteotomy of the first metatarsal for hallux valgus using a low profile plate. Foot Ankle Int. 2009 Oct;30(10):976-80. doi: 10.3113/FAI.2009.0976. PMID 19796591
- [Background] Robinson AH, Limbers JP. Modern concepts in the treatment of hallux valgus. J Bone Joint Surg Br. 2005 Aug;87(8):1038-45. doi: 10.1302/0301-620X.87B8.16467. No abstract available. PMID 16049235
- [Background] Okuda R, Kinoshita M, Yasuda T, Jotoku T, Shima H. Proximal metatarsal osteotomy for hallux valgus: comparison of outcome for moderate and severe deformities. Foot Ankle Int. 2008 Jul;29(7):664-70. doi: 10.3113/FAI.2008.0664. PMID 18785415
- [Background] Thordarson DB, Leventen EO. Hallux valgus correction with proximal metatarsal osteotomy: two-year follow-up. Foot Ankle. 1992 Jul-Aug;13(6):321-6. doi: 10.1177/107110079201300605. PMID 1398360